CLINICAL TRIAL: NCT04418271
Title: Prehabilitation of Elderly Frail or Pre-frail Patients Prior to Elective Surgery - a Randomized Controlled Multicenter Study (PRAEP-Go)
Brief Title: Prehabilitation of Elderly Patients With Frailty Syndrome Before Elective Surgery (PRAEP-GO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Technische Universität Berlin (Other); BARMER (Other)
Responsible Party: Principal Investigator, Claudia Spies, Univ.- Prof. Dr. Claudia Spies, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRAEP-GO; U1111-1253-4820 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2020-05-19; First posted 2020-06-05 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Frailty; Frail Elderly
Keywords: Prehabilitation, Physiotherapy, Exercise Therapy, Rehabilitation, Nutritional Intervention, Multidisciplinary Intervention, Frailty, Surgery
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Patients with frailty syndrome (≥1 of the standardized parameters (Pre-Frail = 1-2; Frail≥3) according to Fried et al.(2001) are offered randomised participation in the new form of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Prefrail and frail patients receive prehabilitation (new form of care)
  Interventions: Behavioral: Prehabilitation- new form of care
- Standard of Care (No Intervention): Prefrail and frail patients receive no prehabilitation, but receive standard of care

INTERVENTIONS:
Behavioral: Prehabilitation- new form of care — The participants in the intervention group take part in a shared decision-making (SDM) conference to plan the intervention. The therapeutic content of the prehabilitation is defined individually for each patient in the SDM conference. Prehabilitation will be a structured and individually tailored 3-week program.
  Arms: Prehabilitation

SUMMARY:
The aim of the study is to evaluate the effect of a shared decision-making conference and three-week prehabilitation program on the outcome "care dependency" one year after surgery. The cost-effectiveness of the intervention will also be evaluated in this N = 1400 patient, national multicenter, assessor-blinded, randomized, pragmatic, controlled, parallel-group, clinical trial.

The objective of PRÄP-GO is to establish and employ a suitable preoperative case-care management system to improve the short and long-term outcome of elderly surgical patients with signs of a frailty syndrome, improving postoperative quality of life and reducing care dependency by a three-week individualized prehabilitation program.

ELIGIBILITY:
Study patients:

Inclusion Criteria:

* Age ≥ 70 years
* Consent by Patient or Legal Representative
* Elective surgery planned
* Expected anesthesia duration≥ 60 min
* Statutory health insurance
* Frailty syndrome (≥1 positive out of 5 standardized parameters according to the Physical Frailty Phenotype according to Fried et. al.)

Exclusion Criteria:

* Severe cardiac or pulmonary disease (NYHA IV, Gold IV)
* Intracranial interventions
* Moribund patients (palliative situation)
* Not enough language skills
* Participation in another interventional rehabilitation study or other interventional clinical trial that has not been approved by the study management committee (Exception: Participation in adjuvant intervention study)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1199 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Degree of care dependency | Up to one year
  Assessment results in a degree of care dependency from personal help according to the German dependency assessment (= "Neues Begutachtungs-Assessment" (NBA)) (Wingenfeld et al., 2008). The results of the assessments ranges between 0 and 100 points, which are transformed into a 0-5 ordinal scale. Higher points in the assessments indicate higher demand of care dependency. Accordingly, higher numbers on the ordinal scale indicate a higher level of care dependency as defined in the German statutory care insurance program.

SECONDARY OUTCOMES:
Barthel Index | Up to one year
  Level of care dependency after surgery reported as Barthel Index
Change in NBA score | Up to one year
  Assessment results according to the German dependency assessment (= "Neues Begutachtungs-Assessment" (NBA)) (Wingenfeld et al., 2008) using the results of the assessments on the scale from 0 to 100 points
NBA domain change | Up to one year
  Change in individual domains of the German dependency assessment (= "Neues Begutachtungs-Assessment" (NBA)).
Surrogate for Neurocognitive Disorder (NCD) | Up to one year
  Frequency of neurocognitive vulnerability at 3 or 12 months as surrogate for NCD is measured as composite score:
  1. Frequency of cognitive impairment/vulnerability is calculated from a change in composite of MiniCog, ANT, TMT-B and MOCA
  2. subjective concern (MMQ) and
  3. IADL/ADL
Screening tool for cognitive vulnerability | Up to one year
  Cognitive vulnerability is suspected by limited MiniCog-test result. The MiniCog consists of two items, the word recall test and the clock-drawing test. Performance in these test is rated on a scale ranging from 0 - 5, with <3 points indicating a cognitive vulnerability.
Dementia risk assessed by MOCA | Up to one year
  Dementia risk is assessed by Montreal Cognitive Assessment (MOCA-30) deterioration (change) and its absolute value if < 26.
Delirium | Up to one year
  Delirium as perioperative complication assessed until hospital discharge using billing data.
Frailty | Up to one year
  Frailty is operationalized using modified Fried frailty criteria. Frailty scores from 0 to 5 (i.e., 1 point for each component; 0 = best to 5 = worst) represent robust (0), pre-frail (1-2), and frail (3-5) health status.
Perioperative complications by Clavien-Dindo | Up to hospital discharge
  Perioperative complications assessed using Clavien Dindo till hospital discharge
Every mobility | Up to one year
  Level of everyday mobility using Life-Space Assessment (LSA)
Autonomy Preference | At the beginning of the observation
  Extent of patients' autonomy preference concerning medical decisions; Autonomy-Preference-Index, modified German version (API-Dm). The scale consists of a 11-item questionnaire with 4 questions on preferred autonomy in health-related decisions and 7 items on information preference. The total results of the API and both subscales are transformed into a 0 - 100 scale with higher values indicating higher levels on autonomy and information preference, respectively.
Extent of involvement in shared decision-making process | At the beginning of the observation
  Extent of patients, relatives and health professionals' involvement in shared decision-making process; 9-Item Shared Decision Making Questionnaire (SDM-Q-9/SDM-Q-Doc)
Arm circumference | Up to one year
  Arm circumference is measured in a standardized position and documented in centimeter.
Calf circumference | Up to one year
  Calf circumference is measured in a standardized position and documented in centimeter.
Nutritional Status | Up to one year
  Changes of nutritional status after elective surgery.
Change in body weight | Up to one year
  Changes in body weight measured in kg.
Instrumental Activities of daily living (IADL) | Up to one year
  Instrumental Activities of daily living (IADL) using the questionnaire by Lawton and Brody.
Functional endurance | Up to one year
  Functional endurance is measured using the 2-Minute-Step-Test (2-MST). The patient steps in place, raising each leg to a marker. The markers height is derived from biometrical measures of the patient. The assessor counts each step of the right leg in which the knee of the patient passes the marker. Higher counts of steps indicates better functional endurance.
Function of the respiratory system | Up to one year
  The function of the respiratory system is assessed by expiratory peak flow measurement as surrogate parameter.
Depression | Up to one year
  Depression is measured by frequency of depressive symptoms; Patient Health Questionnaire-8 (PHQ-8)]
Anxiety | Up to one year
  Anxiety is measured frequency of anxiety symptoms; Generalized Anxiety Disorder Scale-7 (GAD-7)
Health related quality of life | Up to one year
  Health related quality of life is measured with EQ-5D-5L questionnaire.
Disability by WHODAS 2.0 | Up to one year
  Patient- or proxy-reported functioning and disability is measured by the WHO Disability Assessment Schedule (WHODAS 2.0, 12-item version.
Falls | Up to one year
  Incidence of falls
Fear of Falling | Up to one year
  Activities-Specific Balance Confidence (ABC)-6-Scale. The scale consists of 6 questions who are rated on a 0-100 NRS-scale. The total result of the ABC-6-scale comprises of the average of all 6 items.
Satisfaction with the intervention: ZUF-8 | Up to one year
  The satisfaction of the patient is measured with the questionnaire on patient satisfaction (ZUF-8). The ZUF-8 is a questionnaire on patient satisfaction after treatment. It consists of 8 questions which results in a score between 0 and 24 points, with higher values.indicating higher levels of satisfaction.
Mortality | Up to one year
  Data from patient records and residents' registration
Muscle strength | Up to one year
  Muscle strength measured by handgrip strength
Functional mobility | Up to one year
  Functional mobility is measured with gait speed over 15ft
Stair climbing speed | Up to one year
  Stair climbing speed test
Timed Up & Go Test (TUG | Up to one year
  Timed Up & Go Test (TUG) to test mobility and body balance
Postoperative functional mobility | Up to one year
  Postoperative complication of mobilization speed measured with CHARMI
Length of stay Intensive Care Unit | Participants are followed up for the duration of rehabilitation, an expected average of 1 day]
  Intensive care unit length of stay describes every day spent in an ICU bed.
Admission Intensive Care Unit (ICU) Admission rate on Intensive Care Unit (ICU) | Participants are followed up for the duration of rehabilitation, an expected average of 1 day]
  Admission rate (planned / unplanned) on ICU
Duration of hospital stay | Participants are followed up for the duration of rehabilitation, an expected average of 7 days]
  Time in hospital

OTHER OUTCOMES:
Adverse Discharge Disposition | Participants are followed up after hospital discharge for 1 day
  Adverse discharge disposition other than to home and planned rehabilitation facility.
Necessity for follow-up treatment and rehabilitation | Up to one year
  Assessment if a follow-up treatment or rehabilitation is necessary after the hospital stay.
Count of new discharge diagnoses | Participants are followed up for the duration of rehabilitation, an expected average of 7 days]
  New medical diagnoses at hospital discharge compared to baseline are assessed.
Count of new discharge medication | Participants are followed up for the duration of rehabilitation, an expected average of 7 days]
  New medication at hospital discharge compared to baseline is assessed.
Duration of rehabilitation | Participants are followed up for the duration of rehabilitation, an expected average of 25 days]
  Patient record data, discharge letter
Health economic benefit | Up to one year
  ScreeningThe health economic benefit of the intervention (prehabilitation) will be compared to standard of care in the German health care system using a health cost analysis framework.
Exercise adherence and planned prehabilitation composition | Up to one year
  Assessment of the appropriateness of the quantity and quality of the exercise interventions compared to exercise prescription guidelines.
Patient support | Up to one year
  Patient support by need/prescription of assistive devices ("Hilfsmittel") and therapeutic treatment ("Heilmittel").
Polypharmacy | Up to one year
  Measured by number of drug agents
Alcohol Use | Up to one year
  Measured by Alcohol Use Disorders Identification Test (AUDIT-C)
Tobacco Use | Up to one year
  Measured by Fagerstrom (Fagerstrom & Schneider, 1989)
Sarcopenia | Up to one year
  Sarcopenia is evaluated as a composite measure by three criteria that are assessed: 1) low muscle strength (hand grip strength), 2) low muscle quantity (calf circumference) and 3) low physical performance (gait speed or TUG).
Social situation measurement 1 | Up to one year
  The social situation 1 of the patient is measured by a Questionnaire for Social Situation (SOS, Subscales 1 and 2).
Social situation measurement 2 | Up to one year
  The social situation 2 of the patient is measured by BSSS, 8-items
Pain: Numeric rating scale | Up to one year
  Pain is measured with a pain score Numeric rating scale (0-10), a higher score indicates more pain.
Loneliness | Up to one year
  Frequency of sensations of loneliness; 3-item UCLA Loneliness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, Prof., MD, Study Chair — Charite University, Berlin, Germany
Locations (23):
- Germany (23):
  - Herz- und Diabetes Zentrum, Bad Oeynhausen
  - Department of Anesthesiology and Operative Intensive Care Medicine (CBF), Charité - Universitätsmedizin Berlin, Berlin
  - Department of Anesthesiology and Operative Intensive Care Medicine CCM/CVK, Charité - Universitätsmedizin Berlin, Berlin
  - Auguste-Viktoria-Klinikum - Vivantes - Netzwerk für Gesundheit GmbH, Berlin
  - Bundeswehrkrankenhaus, Berlin
  - CARITAS Klinik Maria Heimsuchung, Berlin
  - Dominikus-Krankenhaus, Berlin
  - Evangelisches Krankenhaus Hubertus, Berlin
  - Humboldt-Klinikum - Vivantes - Netzwerk für Gesundheit GmbH, Berlin
  - Klinikum im Friedrichshain - Vivantes - Netzwerk für Gesundheit GmbH, Berlin
  - Martin-Luther-Krankenhaus, Berlin
  - Sankt Joseph Krankenhaus, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Klinikum Frankfurt Oder GmbH, Frankfurt (Oder)
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Sana Kliniken Sommerfeld, Kremmen
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Universität zu Lübeck, Lübeck
  - Klinikum der Universität München, LMU Campus Großhadern, München
  - Klinikum rechts der Isar - Technische Universität München, München
  - München Klinik Bogenhausen, München
  - Havelland Kliniken GmbH - Klinik Nauen, Nauen
  - Havelland Kliniken-Klinik Rathenow, Rathenow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schone C, Fuchs TI, Kiselev J, Schmidt K, Schaller SJ, Spies C, Rombey T. Facilitators and barriers to participation in prehabilitation prior to orthopaedic elective surgery - a qualitative study with elderly (pre-)frail patients. BMC Geriatr. 2025 Nov 4;25(1):845. doi: 10.1186/s12877-025-06592-3. PMID 41188708
- [Derived] Eckhardt H, Quentin W, Silzle J, Busse R, Rombey T. Cost-effectiveness of prehabilitation of elderly frail or pre-frail patients prior to elective surgery (PRAEP-GO) versus usual care - Protocol for a health economic evaluation alongside a randomized controlled trial. BMC Geriatr. 2024 Mar 6;24(1):231. doi: 10.1186/s12877-024-04833-5. PMID 38448804
- [Derived] Schaller SJ, Kiselev J, Loidl V, Quentin W, Schmidt K, Morgeli R, Rombey T, Busse R, Mansmann U, Spies C; PRAEP-GO consortium,; PRAEP-GO investigators. Prehabilitation of elderly frail or pre-frail patients prior to elective surgery (PRAEP-GO): study protocol for a randomized, controlled, outcome assessor-blinded trial. Trials. 2022 Jun 6;23(1):468. doi: 10.1186/s13063-022-06401-x. PMID 35668532